CLINICAL TRIAL: NCT05180539
Title: A Multi-Component Alcohol and Sex Risk Intervention for College Students
Acronym: SPLASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh University (Other)
Collaborators: Brown University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Interventional; 5R34AA026032 (NIH)
Record Dates: First submitted 2021-09-09; First posted 2022-01-06 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: College Drinking
MeSH Terms: conditions — Alcohol Drinking in College

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPLASH Intervention Condition (Experimental): Two in-person group sessions addressing alcohol harm reduction and intervening to reduce sexual violence in drinking contexts
  Interventions: Behavioral: SPLASH Intervention Condition
- Diet and Physical Activity Condition (Other): Two in-person group sessions addressing increasing healthy eating and physical activity
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: SPLASH Intervention Condition — Two-session in person group discussions focusing on behaviors in drinking contexts
  Arms: SPLASH Intervention Condition
Behavioral: Control Condition — Two-session in person group discussions focusing on college health behaviors
  Arms: Diet and Physical Activity Condition

SUMMARY:
Hazardous alcohol use, sexually transmitted infections, and sexual violence are interrelated and highly prevalent public health concerns in college student populations. The current study seeks to develop a tri-pronged sex-positive intervention that addresses risky alcohol use, unsafe sex, and sexual violence for college men and women (ages 18-24). The study involves a small randomized pilot trial to demonstrate the feasibility and acceptability of the recruitment methods and research design. Preliminary evidence of intervention efficacy will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Must be student at the site university

Exclusion Criteria:

* Students who have participated in relevant site specific studies will be excluded

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 274 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Napper, PhD, Principal Investigator — Lehigh University; Shannon Kenney, PhD, Principal Investigator — Brown University
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial recruitment occurred between 9/23/21 and 10/12/21 at two U.S. colleges
Pre-assignment Details: Participants who consented to participate were not assigned to condition if: (1) they were unavailable to attend intervention meetings, (2) they expressed they were no longer interested in participating after completing baseline assessment, or (3) they withdrew for unknown reasons prior to randomization (e.g., they did not complete information necessary to sign up to attend the intervention sessions).
Period: Overall Study
Arm/Group | SPLASH Intervention Condition | Diet and Physical Activity Condition
Started | 134 | 140
Completed (If participants missed a data collection point, they were still able to complete later data collection timepoints. These numbers reflect the total number participants in each condition who met the criteria to be included in the analyses, not the number who complete the final data collection timepoint.) | 107 | 110
Not Completed | 27 | 30
Not completed — Lost to Follow-up | 27 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPLASH Intervention Condition | Diet and Physical Activity Condition | Total
Number analyzed (Participants) | 134 | 140 | 274
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 134 | 140 | 274
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 64 | 58 | 122
  Male | 68 | 76 | 144
  Transgender/non-binary | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 20 | 46
  Not Hispanic or Latino | 108 | 120 | 228
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 34 | 28 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 12 | 18
  White | 78 | 85 | 163
  More than one race | 13 | 12 | 25
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 134 | 140 | 274
Drank alcohol past 30 days [Count of Participants; unit: Participants] | 87 | 94 | 181
Had unprotected sex past 30 days [Count of Participants; unit: Participants] | 36 | 41 | 77

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome: Program Satisfaction as Assessed by the Acceptance Questionnaire After First Intervention Session
Description: Satisfaction with the program content after Session 1. Percent of participants reporting they were moderately-to-very satisfied with the program.
Time Frame: Immediate post intervention (same day as intervention), after first session on day 1
Population: Program satisfaction not examined in control condition (diet and physical activity group). Missing data reflects the study design. Participants could attend 1 or 2 study sessions. Data is missing for participants who did not attend the first in-person session (follow-up data was still collected for these participants).
Measure: Count of Participants; unit: Participants
Arm/Group | SPLASH Intervention Condition
Number analyzed (Participants) | 99
Participants
  Overall Satisfaction (after Session 1) | 86
  Would recommend program to friend (after Session 1) | 91

2. Primary Outcome: Program Satisfaction as Assessed by the Acceptance Questionnaire After Second Session
Description: Satisfaction with the program content after session 2. Percent of participants reporting that they were moderately-to-very satisfied with the program. For participants who did not attend the first session this occurred on Day 1. For Participants who did attend the first session this occurred around Day 14 (range between day 12 and 17)
Time Frame: Immediate post intervention (same day as intervention), after second session on ~Day 14
Population: Program satisfaction not examined in control condition (diet and physical activity group). Missing data reflects the study design. Participants could attend 1 or 2 study sessions. Data is missing for participants who did not attend the second in-person session (follow-up data was still collected for these participants).
Measure: Count of Participants; unit: Participants
Arm/Group | SPLASH Intervention Condition
Number analyzed (Participants) | 87
Participants
  Overall Satisfaction (After Session 2 [~ Day 14) | 83
  Would recommend program to friend (After Session 2) [~ Day 14): number analyzed (Participants) | 86
  Would recommend program to friend (After Session 2) [~ Day 14) | 83

3. Primary Outcome: Heavy Alcohol Use
Description: Number of standard drinks consumed in a typical week over the past 30 days
Time Frame: Change from baseline to 6 month follow-up
Population: Participants who did not complete the 1 month follow up survey were still able to complete the 6 month follow up survey. The analysis sample reflects participants who completed the baseline survey, attended at least 1 in-person group meeting, and completed at least one follow up survey (1 month or 6 month). Adjusted means are reported from a Generalized Estimating Equations (GEE) model that accounts for missing data if participants missed a follow-up survey.
Measure: Mean (Standard Error); unit: Drinks per week
Arm/Group | SPLASH Intervention Condition | Diet and Physical Activity Condition
Number analyzed (Participants) | 106 | 109
Drinks per week
  Baseline | 7.1 (0.8) | 5.6 (0.7)
  1 month | 6.7 (0.7) | 5.3 (0.6)
  6 months | 6.0 (0.7) | 4.7 (0.6)

4. Primary Outcome: Alcohol Use Before or During Sex
Description: Participants reported if they drank alcohol before or during sex in the past 30 days (code as yes = 1 or no = 0).
Time Frame: Change from baseline to 6 month follow-up
Population: Participants who did not complete the 1 month follow up survey were still able to complete the 6 month follow up survey. The analysis sample reflects participants who completed the baseline survey, attended at least 1 in-person group meeting, and completed at least one follow up survey (1 month or 6 month). Adjusted proportions are reported from a GEE model that accounts for missing data if participants missed a follow-up survey.
Measure: Number; unit: adjusted percentage of participants
Arm/Group | SPLASH Intervention Condition | Diet and Physical Activity Condition
Number analyzed (Participants) | 107 | 110
adjusted percentage of participants
  Baseline | 0.3 | 0.3
  1 month | 0.4 | 0.4
  6 months | 0.3 | 0.3

5. Primary Outcome: Bystander Behaviors Willingness Questionnaire
Description: Willingness to engage in bystander behaviors. Mean scale scores range from 1 to 7. Higher scores indicate more greater willingness to engage in bystander behaviors.
Time Frame: Change from baseline to 6 month follow-up
Population: Participants who did not complete the 1 month follow up survey were still able to complete the 6 month follow up survey. The analysis sample reflects participants who completed the baseline survey, attended at least 1 in-person group meeting, and completed at least one follow up survey (1 month or 6 month). Adjusted means are reported from a mixed model that accounts for missing data if participants missed a follow-up survey.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | SPLASH Intervention Condition | Diet and Physical Activity Condition
Number analyzed (Participants) | 106 | 109
Units on a scale
  Baseline | 6.0 (0.1) | 5.8 (0.1)
  1month | 5.1 (0.1) | 5.1 (0.1)
  6months | 6.0 (0.1) | 5.9 (0.1)

6. Primary Outcome: Bystander Behaviors Self-efficacy Questionnaire
Description: Confidence to engage in bystander behaviors. Higher scores indicate more greater confidence in ability to engage in bystander behaviors. Mean scale scores range from 1 to 5.
Time Frame: Change from baseline to 6 month follow-up
Population: Participants who did not complete the 1 month follow up survey were still able to complete the 6 month follow up survey. The analysis sample reflects participants who completed the baseline survey, attended at least 1 in-person group meeting, and completed at least one follow up survey (1 month or 6 month). Adjusted means are reported from a GEE model that accounts for missing data if participants missed a follow-up survey.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | SPLASH Intervention Condition | Diet and Physical Activity Condition
Number analyzed (Participants) | 106 | 109
units on a scale
  Baseline | 4.1 (.07) | 4.0 (.07)
  1 month | 4.0 (.09) | 4.1 (.09)
  6 months | 4.1 (.09) | 3.9 (.08)

7. Secondary Outcome: Alcohol and Sex Related Protective Behavioral Strategies Use
Description: Self-reported frequency of using strategies to reduce alcohol risks and promote positive sexual experiences [unpublished measure]. Higher scores indicate more frequent use of protective strategies. Scores range from 0 to 5 for both subscales.
Time Frame: Change from baseline to 6 month follow-up
Population: Strategies related to drinking were analyzed separately to those related to sex. Participants who did not complete the 1 month follow up survey were still able to complete the 6 month follow up survey. The analysis sample reflects participants who completed the baseline survey, attended at least 1 in-person group meeting, and completed at least one follow up survey (1 month or 6 month). Adjusted means are reported from a mixed model addressing missing data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SPLASH Intervention Condition | Diet and Physical Activity Condition
Number analyzed (Participants) | 103 | 102
score on a scale
  Drinking PBS | 3.4 (.10) | 3.4 (.09)
  Drinking PBS 1 month | 3.6 (0.12) | 3.3 (.11)
  Drinking PBS 6 months | 3.5 (0.12) | 3.5 (.12)
  Sex PBS Baseline: number analyzed (Participants) | 103 | 100
  Sex PBS Baseline | 3.4 (.13) | 3.2 (.12)
  Sex PBS 1 month | 3.3 (0.15) | 3.3 (.15)
  Sex PBS 6 months | 3.7 (.15) | 3.4 (.14)

8. Secondary Outcome: Perceived Student Drinking Norms as Assessed by the Drinking Norms Rating Form
Description: Perceived descriptive norms are assessed using a variation on the Drinking Norms Rating Form. Respondents estimate the number of standard drinks consumed by other students on their campus for each day in a typical week in the past 30 days; daily estimates are summed to yield perceived number of drinks per week for student peers; range of scores can go from zero to no upper limit
Time Frame: Change from baseline to 6 month follow-up
Population: Adjusted means are reported from a Generalized Estimating Equations (GEE) model addressing missing data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SPLASH Intervention Condition | Diet and Physical Activity Condition
Number analyzed (Participants) | 106 | 108
score on a scale
  Baseline | 13.1 (.9) | 13.5 (.9)
  1 month | 10.1 (.7) | 10.8 (.7)
  6 months | 10.4 (.7) | 13.0 (.7)

9. Secondary Outcome: Perceived Student Sex Norms as Assessed by a Sex Norms Questionnaire
Description: Respondents estimate the percent of same-campus peers who use alcohol before or during sex
Time Frame: Change from baseline to 6 month follow-up
Population: Adjusted means are reported from a mixed model addressing missing data.
Measure: Mean (Standard Error); unit: perceived percentage of other students
Arm/Group | SPLASH Intervention Condition | Diet and Physical Activity Condition
Number analyzed (Participants) | 99 | 94
perceived percentage of other students
  Baseline Norms | 54.6 (2.4) | 56.0 (2.3)
  1 month norms | 36.7 (2.5) | 52.9 (2.5)
  6 month norms | 44.1 (2.6) | 54.0 (2.4)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | SPLASH Intervention Condition | Diet and Physical Activity Condition
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/110
Other Adverse Events (participants affected / at risk) | 0/107 | 0/110

LIMITATIONS AND CAVEATS:
Trial was primarily designed to test feasibility and acceptability and not powered sufficiently to detect group differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT05180539/Prot_SAP_000.pdf